CLINICAL TRIAL: NCT03593317
Title: Blockade of the Renin-angiotensin-aldosterone System in Patients With ARVD: a Double-blind Multicentre Prospective Randomized Study.
Brief Title: Blockade of the Renin-angiotensin-aldosterone System in Patients With ARVD
Acronym: BRAVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL18_0038; 2023-505048-20-00 (Other: EUCT)
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Arrhythmogenic Right Ventricular Dysplasia
Keywords: Heart Failure; Right ventricle
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Heart Failure | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spironolactone group (Experimental)
  Interventions: Drug: Spironolactone
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — The doses used in the study are the doses used in standard clinical practice. Initial dose is 25 mg/day until study end . The duration of treatment for each patient is 12 months.
  Arms: Spironolactone group
Drug: Placebo — Placebo will be taken once a day at the same time of day. The duration of treatment for each patient is 12 months.
  Arms: Placebo group

SUMMARY:
Arrhythmogenic right ventricular dysplasia (ARVD) is a rare cardiomyopathy characterized by the progressive replacement of cardiomyocytes by fatty and fibrous tissue in the right ventricle (RV). These infiltrations lead to cardiac electrical instability and ventricular arrhythmia.

Current treatment for ARVD is empirical and essentially based on treatment of arrhythmia. Thus, there is no validated treatment that will prevent the deterioration of the RV function in patients with ARVD.

The investigator's hypothesis is that the use of anti-fibrotic medications will prevent or at least reduce the deterioration of the RV function. The aim of this project is to evaluate the effect of spironolactone, a Potassium-sparing diuretic on ventricular myocardial remodeling and on arrhythmia burden in patients with ARVD.

The trial is a double-blind parallel multicenter prospective randomized phase II drug study. Patients will be randomized in the two groups: spironolactone or placebo. 13 centers in France will enroll the 120 patients (60 per group). Patients will be followed for 3 years (6 months, 1 year and 3 years) with all examinations (ECG, HA ECG, 24-hour Holter, trans-thoraciqc echocardiography (TTE), biological analyses) according to standard of care. A decrease in right and/or left ventricular deterioration and in arrhythmia burden are expected in ARVD patients treated with spironolactone. This reduction will improve the quality of life of patients and will reduce the number of hospitalizations and the risk of terminal heart failure.

ELIGIBILITY:
Inclusion Criteria:

* >18years old
* Diagnosis of ARVD based on Task Force criteria. Two major criteria: 1 morphologic and one rhythmic or 1 major and 2 minor criteria established by the European Society of Cardiology/International Society and Federation of Cardiology.
* Left Ventricular Ejection Fraction >40%
* Written informed consent.

Exclusion Criteria:

* Patients under judicial protection.
* Female patient who is pregnant or lactating, or is of child bearing potential (defined as a sexually mature woman not surgically sterilized or not post-menopausal for at least 24 consecutive months if ≤ 55 years or 12 months if > 55 years) and who did not agree to use highly effective methods of birth control throughout the study.
* No health insurance.
* Right heart failure patient (RV volume>150ml).
* Spironolactone contraindication: anuria, hyperkalemia (K+>5 mmol/l), renal failure (DFGCréat>22 mL/min/1,73 m2), end-stage liver failure, Addison's Disease, hypersensitivity to spironolactone or to any of the excipients (patients with galactose intolerance, lapp lactase deficiency or glucose or galactose malabsorption syndrome), association with eplerenone, association with other hyperkalemic diuretics, association with potassium salts, not recommended in cirrhotic patients (natraemia<125 mmol/l) or in patients likely to present an acidosis.
* Mandatory indication for a combination of ACE inhibitor and sartan or renin inhibitor (each authorized separately).
* Acute phase of systemic disease.
* Uncompensated hypothyroidism.
* Acute hyperthyroidism.
* Normal right ventricular volume.
* Heart transplantation.
* Swallowing disorders.
* Participation in any other interventional clinical investigation that may have an impact on our study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Right ventricle longitudinal strain measured by echocardiography | at year 1
Right ventricle infundibulum diameter measured by echocardiography | at year 1
number of ventricular extrasystoles > 500 on 24h-Holter ECG | at year 1

SECONDARY OUTCOMES:
number of ventricular extrasystoles on 24h-Holter ECG | at year 1
number of palpitations | at year 1
number of palpitations | at year 3
number of ventricular tachycardia | at year 1
number of ventricular tachycardia | at year 3
number of dyspnea | at year 1
number of dyspnea | at year 3
number of syncope | at year 1
number of syncope | at year 3
number of sudden death | at year 1
number of sudden death | at year 3
number of thoracic pain | at year 1
number of thoracic pain | at year 3
number of MACE (Major adverse cardiac events) | at year 1
number of MACE (Major adverse cardiac events) | at year 3
number of hospital admissions | at year 1
number of hospital admissions | at year 3
left ventricle diameters measured by echocardiography | at year 1
  Morphologic criterion
left ventricle diameters measured by echocardiography | at year 3
  Morphologic criterion
left ventricle volumes measured by echocardiography | at year 1
  Morphologic criterion
left ventricle volumes measured by echocardiography | at year 3
  Morphologic criterion
left ventricle ejection fraction measured by echocardiography | at year 1
  Morphologic criterion
left ventricle ejection fraction measured by echocardiography | at year 3
  Morphologic criterion
Left ventricular global longitudinal strain measured by echocardiography | at year 1
  Morphologic criterion
aneurism measured by echocardiography | at year 1
  Morphologic criterion
aneurism measured by echocardiography | at year 3
  Morphologic criterion
dyskinesia measured by echocardiography | at year 1
  Morphologic criterion
dyskinesia measured by echocardiography | at year 3
  Morphologic criterion
evolution of QRS width (50mm/s) on ECG | at year 1
  Morphologic criterion
number of ventricular extrasystoles on 24h Holter ECG | at year 1
  Rhythmic criterion
sustained ventricular tachycardia on 24h Holter ECG | at year 1
  Rhythmic criterion
evolution of PR interval duration on ECG | at year 1
  Rhythmic criterion
late potentials measured with high amplification ECG | at year 3
  Rhythmic criterion
number of ventricular extrasystoles by stress test | at year 3
  Rhythmic criterion
Evolution of functional symptoms by recording adverse events | at year 3
  Functional criteria
Number of hospital admissions owing to clinical deterioration | at year 3
Evolution of telediastolic right ventricle volume measured by echocardiography | at year 3
  according to the genotype of desmosome genes
arrhythmia burden measured by 24h Holter ECG | at year 3
  according to the genotype of desmosome genes
Dosage of MMP9 (Matrix metallopeptidase 9) | at year 1
  Quantification of fibrosis
Dosage of MMP9 (Matrix metallopeptidase 9) | at year 3
  Quantification of fibrosis
Dosage of TIMP1 (Tissue Inhibitory MetalloProtease 1) | at year 1
  Quantification of fibrosis
Dosage of TIMP1 (Tissue Inhibitory MetalloProtease 1) | at year 3
  Quantification of fibrosis
Dosage of TIMP2 (Tissue Inhibitory MetalloProtease 2) | at year 1
  Quantification of fibrosis
Dosage of TIMP2 (Tissue Inhibitory MetalloProtease 2) | at year 3
  Quantification of fibrosis
Dosage of IL6 (Interleukin 6) | at year 1
  Quantification of inflammation
Dosage of IL6 (Interleukin 6) | at year 3
  Quantification of inflammation
Dosage of IL8 (Interleukin 8) | at year 1
  Quantification of inflammation
Dosage of IL8 (Interleukin 8) | at year 3
  Quantification of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Chevalier, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (13):
- France (13):
  - CHU Amiens Picardie, Amiens
  - Hôpital Cardiologique Louis Pradel, Bron
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU Dijon, Dijon
  - Hôpital Michallon, Grenoble
  - Hôpital de la Timone, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital Laennec, Nantes
  - Groupe Hospitalo Universitaire Caremeau, Nîmes
  - Hôpital Pitié Salpetrière, Paris
  - Hôpital de Haut-Lévêque, Pessac
  - Nouvel Hôpital Civil, Strasbourg
  - Hôpital Rangueil, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided